CLINICAL TRIAL: NCT04395170
Title: A Randomized, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of the Use of Convalescent Plasma (PC) and Human Intravenous Anti COVID-19 Immunoglobulin (IV Anti COVID-19 IgG) in Patients Hospitalized for COVID-19.
Brief Title: Convalescent Plasma (PC) and Human Intravenous Anti-COVID-19 Immunoglobulin (IV Anti COVID-19 IgG) in Patients Hospitalized for COVID-19.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lifefactors Zona Franca, SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LFCOLCOVID-19-001
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — COVID-19 Serotherapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Convalescent plasma (Experimental): Plasma from patients recovering from COVID-19.
  Interventions: Biological: COVID-19 convalescent plasma
- Anti-COVID-19 human immunoglobulin (Experimental): Anti-COVID-19 human immunoglobulin to be administered intravenously.
  Interventions: Biological: Anti-COVID-19 human immunoglobulin
- Standard (specific) therapy (Active Comparator): Standard therapy for COVID-19 according to the recommended pharmacological recommendations of the Colombian Association of Infectious Diseases - ACIN. This therapy is subject to changes that are defined by the Colombian Health Regulatory Authorities.
  To date, these therapies may include remdesivir, chloroquine, hydroxychloroquine, azithromycin.
  Interventions: Drug: Standard (specific) therapy for COVID-19

INTERVENTIONS:
Biological: COVID-19 convalescent plasma — Plasma from convalescent patients with COVID-19 and at the same time receiving supportive therapy, with inactivation / reduction of pathogens, in the scheme of two doses of 200 - 250 mL administered on days 1 and 3 of the intervention.
  Arms: Convalescent plasma
Biological: Anti-COVID-19 human immunoglobulin — Anti-COVID-19 human immunoglobulin produced by Lifefactors Zona Franca S.A.S, intravenously at a dose of immunoglobulin 10% IgG solution (10% mL vial) for:
  Patient of 50 Kg or more, a dose of 50 mL, administered on days 1 and 3 of treatment.
  Patient under 50 Kg, the dose will be 1 mL / Kg, administered on days 1 and 3 of treatment.
  The supply of anti-COVID-19 human immunoglobulin produced by Lifefactors Zona Franca S.A.S included once it has been authorized by INVIMA and/or the regulatory requirements in force for the production of drugs are met.
  Arms: Anti-COVID-19 human immunoglobulin
Drug: Standard (specific) therapy for COVID-19 — Standard therapy for COVID-19 according to the recommended pharmacological recommendations of the Colombian Association of Infectious Diseases - ACIN. This therapy is subject to changes that are defined by the Colombian Health Regulatory Authorities.
  To date, these therapies may include remdesivir, chloroquine, hydroxychloroquine, azithromycin.
  Arms: Standard (specific) therapy

SUMMARY:
A randomized, open-label, multicenter, three-arm clinical trial to study the efficacy and safety of passive immunotherapy (convalescent plasma and anti-COVID-19 human immunoglobulin) compared to the standard treatment in Colombia.

DETAILED DESCRIPTION:
The study population will be patients (≥18 years) hospitalized by COVID-19 but still with an early form of the disease (in states 1-3 of the ordinal scale) who do not require mechanical ventilation (invasive or non-invasive) and who can give their consent informed.

All the participants will receive non-specific supportive treatment for COVID-19 such as oxygen, IV liquid or corticosteroids. Additionally, they will be randomized to one of the following arms:

Experimental arm 1: Plasma with inactivation/reduction of pathogens from convalescent patients with COVID-19 and who at the same time receive support therapy, in the 200 - 250 mL scheme, on days 1 and 3 of the intervention.

Experimental arm: Anti-COVID-19 human immunoglobulin produced by Lifefactors Zona Franca S.A.S, intravenous at a dose of immunoglobulin 10% IgG solution (10% mL vial) for:

Patient of 50 Kg or more, a dose of 50 mL will be applied on days 1 and 3 of treatment.

Patients of less than 50 Kg, the dose will be 1 mL / Kg, will be applied on days 1 and 3 of treatment.

This arm will be included once available. The supply of anti-COVID-19 human immunoglobulin produced by LifeFactors will be carried out once the national regulatory agency (Invima) grants authorization and/or the regulatory requirements for the production of medications are met.

Control arm: Standard (specific) therapy for COVID-19 according to the suggested pharmacological recommendations of the Colombian Association of Infectious Diseases - ACIN. This therapy is subject to changes that are determined by the Colombian Health Regulatory Authorities.

ELIGIBILITY:
Inclusion Criteria:

1. Obtaining the informed written consent before carrying out the study procedures, by the patients.
2. Adult patients ≥18 years at the time of recruitment for the study.
3. Patients with laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction on nasal/oropharyngeal swabs or any other relevant specimen <72 hours before randomization.
4. Patients requiring hospitalization for COVID-19 without mechanical ventilation (invasive or non-invasive, including an oxygen mask with reserve bag) and at least one of the following:

   1. Radiographic evidence of pulmonary infiltrates by images (chest radiography, computed tomography, etc.),
   2. Clinical evaluation (evidence of rales/crackles on examination) and oxygen saturation ≤ 94% in ambient air requiring supplemental oxygen.
5. Patient with no more than 72 hours (3 days) of hospitalization prior to the administration of PC treatment (except the days after initial hospital admission for other reasons and prior to COVID-19 infection).
6. Patients who do not have more than 10 days between the onset of symptoms (fever or cough) and the day of administration of treatment or the demonstration of the absence of anti-SARS-CoV-2 antibodies (patients with more than 10 days of symptoms they can only be included if a negative antibody result has been confirmed).

Exclusion Criteria:

1. Patient in a state of pregnancy.
2. Require mechanical ventilation (invasive or non-invasive, including oxygen mask with reserve bag) on examination.
3. Participation in any other clinical trial of an experimental treatment for COVID-19.
4. At the discretion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, regardless of the provision of treatments.
5. Any incompatibility or allergy to the administration of plasma of human origin.
6. Severe chronic kidney disease in stage 4 or requiring dialysis (that is, glomerular filtration rate <30).
7. Any condition that in the investigator's opinion limits participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Admission to ICU and/or mechanical ventilation | One year
  Admission to the intensive care unit with the requirement of mechanical ventilation (invasive or non-invasive) due to Acute Respiratory Distress Syndrome by COVID-19.

SECONDARY OUTCOMES:
Length of hospital stay | One year
  Time in the hospital from admission to discharge or death.
Neutralizing antibody (IgG) titers against COVID-19 | One year
  Neutralizing antibody (IgG) titers against COVID-19
Safety - Adverse events | One year
  Non-serious adverse events (NSAEs) and serious adverse events (SAEs)
Death | One year
  Overall mortality

CONTACTS AND LOCATIONS:
Locations (1):
- LifeFactors Zona Franca SAS, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No
No.

REFERENCES:
- [Background] Cancer Institute N. Common Terminology Criteria for Adverse Events (CTCAE) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 [Internet]. 2017. Available from: https://www.meddra.org/
- [Result] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Result] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Result] Soo YO, Cheng Y, Wong R, Hui DS, Lee CK, Tsang KK, Ng MH, Chan P, Cheng G, Sung JJ. Retrospective comparison of convalescent plasma with continuing high-dose methylprednisolone treatment in SARS patients. Clin Microbiol Infect. 2004 Jul;10(7):676-8. doi: 10.1111/j.1469-0691.2004.00956.x. PMID 15214887
- [Result] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Result] Francis F, Hall M, Surg, Gaines A. Early use of convalescent serum in influenza. Mil Surg. 1920;47:177-9.
- [Result] rice H, Genereux M, Sinclair C. Hyperimmune Immunoglobulin G. In: Production of Plasma Proteins for Therapeutic Use [Internet]. Hoboken, NJ, USA: John Wiley & Sons, Inc.; 2012.
- [Result] Vargas M, Segura A, Wu YW, Herrera M, Chou ML, Villalta M, Leon G, Burnouf T. Human plasma-derived immunoglobulin G fractionated by an aqueous two-phase system, caprylic acid precipitation, and membrane chromatography has a high purity level and is free of detectable in vitro thrombogenic activity. Vox Sang. 2015 Feb;108(2):169-77. doi: 10.1111/vox.12209. Epub 2014 Dec 3. PMID 25469648
- [Result] Redden WR. Treatment of Influenza-Pneumonia by Use of Convalescent Human Serum. Bost Med Surg J. 1919 Dec 11;181(24):688-91.
- [Result] Wong VW, Dai D, Wu AK, Sung JJ. Treatment of severe acute respiratory syndrome with convalescent plasma. Hong Kong Med J. 2003 Jun;9(3):199-201. PMID 12777656
- [Result] van Griensven J, Edwards T, Baize S; Ebola-Tx Consortium. Efficacy of Convalescent Plasma in Relation to Dose of Ebola Virus Antibodies. N Engl J Med. 2016 Dec 8;375(23):2307-2309. doi: 10.1056/NEJMc1609116. Epub 2016 Nov 14. No abstract available. PMID 27959686
- [Result] Zingher A, Mortimer P. Convalescent whole blood, plasma and serum in the prophylaxis of measles: JAMA, 12 April, 1926; 1180-1187. Rev Med Virol. 2005 Nov-Dec;15(6):407-18; discussion 418-21. doi: 10.1002/rmv.480. No abstract available. PMID 16211552
- [Result] Use of Convalescent Whole Blood or Plasma Collected from Patients Recovered from Ebola Virus Disease for Transfusion, as an Empirical Treatment during Outbreaks Interim Guidance for National Health Authorities and Blood Transfusion Services Use of Convale. 2014.
- [Result] FDA Guidance on Conduct of Clinical Trials of Medical Products during COVID-19 Public Health Emergency | FDA [Internet]. Available from: https://www.fda.gov/regulatory-information/search-fda-guidance-documents/fda-guidance-conduct-clinical-trials-medical-products-during-covid-19-public-health-emergency